CLINICAL TRIAL: NCT01449643
Title: The Influence of Inspiratory Muscular Training on Diaphragmatic Mobility, Lung Function and Quality of Life in Obese Individuals
Brief Title: The Influence of Inspiratory Muscular Training (IMT) on Diaphragmatic Mobility in Morbidly Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Lui-s Henrique Sarmento Tenorio, Master's Degree Student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAAE-0280.0.172.000-10
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: Obesity; Diaphragm; Inspiratory muscular training
MeSH Terms: conditions — Obesity | interventions — Speech Reception Threshold Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT Group (Active Comparator): Threshold IMT provides consistent and specific pressure for inspiratory muscle strength and endurance training, regardless of how quickly or slowly patients breathe. This device incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting (in cm H20). When patients inhale through Threshold IMT, a spring-loaded valve provides a resistance that exercises respiratory muscles through conditioning.
  Interventions: Device: Threshold
- Sham Group (Sham Comparator): Non-training protocol
  Interventions: Device: Sham Threshold

INTERVENTIONS:
Device: Threshold
  Arms: IMT Group
Device: Sham Threshold
  Arms: Sham Group

SUMMARY:
The purpose of this study is whether an inspiratory muscle training protocol would be associated with an improvement in of the diaphragm mobility, an increase in pulmonary function values , gain strength and endurance of respiratory muscles and improving quality of life.

DETAILED DESCRIPTION:
Few studies have investigated the effects of an inspiratory muscle training in obese patients on the diaphragmatic mobility and thickness. Obesity, especially morbid, triggers changes in the respiratory system, which can affect the work activities and daily life of individuals with this multifactorial syndrome. These functional changes in mechanical ventilation may be linked to weakness and poor respiratory muscle strength, so by promoting rehabilitation of these muscles can minimize the losses that come with obesity

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 kg/m²
* Absence of acute or chronic lung disease

Exclusion Criteria:

* Acute or chronic inflammatory process
* Thyroid disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Ultrasound evaluation of the diaphragm mobility | 3 months
  Compare and correlate diapgragm excursion with pulmonary function.

SECONDARY OUTCOMES:
Pulmonary function test | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria S Brasileiro-Santos, D.Sc, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Tenorio LH, Santos AC, Camara Neto JB, Amaral FJ, Passos VM, Lima AM, Brasileiro-Santos Mdo S. The influence of inspiratory muscle training on diaphragmatic mobility, pulmonary function and maximum respiratory pressures in morbidly obese individuals: a pilot study. Disabil Rehabil. 2013;35(22):1915-20. doi: 10.3109/09638288.2013.769635. Epub 2013 May 7. PMID 23651130